CLINICAL TRIAL: NCT04890561
Title: An Open-label, Single Dose Study to Evaluate Lemborexant in Milk of Healthy Lactating Women
Brief Title: A Study to Evaluate Lemborexant in Milk of Healthy Lactating Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2006-A001-010
Record Dates: First submitted 2021-05-13; First posted 2021-05-18 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — lemborexant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lemborexant 10 mg (Experimental): Participants will receive a single dose of lemborexant 10 mg tablet, orally on Day 1.
  Interventions: Drug: Lemborexant

INTERVENTIONS:
Drug: Lemborexant — Lemborexant oral tablets.
  Other Names: E2006; Dayvigo

SUMMARY:
The primary purpose of the study is to estimate the cumulative amount of lemborexant excreted in breast milk following a single dose administration of lemborexant 10 milligram (mg) to healthy lactating women and to estimate the relative infant dose (RID) expressed as a percent of the daily maternal dose.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy lactating female at least 18 years of age and willing to sign an informed consent prior to any study-related activities.
2. The participant must have had a normal term pregnancy and has been actively breastfeeding or pumping for at least 5 weeks postpartum; lactation must be well-established and the mother not experiencing problems with feeding her infant breast milk. Participants planning on weaning their infants independent of study participation, who meet aforementioned requirements, will be considered for enrolment in the study.
3. Is willing not to breastfeed for 11 days after the study drug administration.
4. Breastfeeds an infant who is already able to feed from a bottle.
5. Agrees to collect all breast milk from predose to end of the study using an electric pump provided by the sponsor.
6. Is considered reliable and capable of adhering to the protocol and visit schedule according to the judgment of the investigator.

Exclusion Criteria:

1. Has a positive pregnancy test at Screening or Baseline.
2. Evidence of disease that may influence the outcome of the study within 4 weeks before dosing; example, psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system, or participants who have a congenital abnormality in metabolism.
3. Any history of gastrointestinal surgery that may affect pharmacokinetic (PK) profiles, example, hepatectomy, nephrectomy, digestive organ resection (but not cholecystectomy) at Screening or Baseline.
4. Any clinically abnormal symptom or organ impairment found by medical history at Screening, and physical examinations, vital signs, ECG finding, or laboratory test results that require medical treatment at Screening or Baseline.
5. A prolonged QT interval by Fridericia (QTcF) (QTcF greater than [>] 450 milliseconds [ms]) as demonstrated by a repeated ECG at Screening.
6. Any suicidal behavior (per the Suicidal Behavior section of the Columbia-Suicide Severity Rating Scale) within 10 years of Screening.
7. Evidence of clinically significant disease (example, cardiac, respiratory, gastrointestinal, renal disease) that in the opinion of the investigator(s) could affect the participant's safety or interfere with the study assessments.
8. Exposure within the last 14 days to an individual with confirmed or probable coronavirus disease (COVID-19) or symptoms within the last 14 days that are on the most recent centers for disease control and prevention (CDC) list of COVID symptoms or any other reason to consider the participant at potential risk for an acute COVID-19 infection.
9. Has mastitis or other condition that would prevent the collection of milk from one or both breasts.
10. Is a smoker (>5 cigarettes, or nicotine equivalent, per day).
11. Has a positive result for urine drug screening.
12. Has undergone surgery (other than caesarean section) or donated blood within 8 weeks prior to the start of the study.
13. Used any prescription or over-the-counter medications, which may impact plasma concentration of lemborexant, within 1 week or 5 half-lives, whichever is longer, before Screening.
14. Hypersensitivity to the study drug or any of the excipients.
15. History of or has concomitant medical condition(s) that in the opinion of the investigator(s) would compromise the participant's ability to safely complete the study.
16. History of drug or alcohol dependency or abuse within approximately the last 2 years.
17. Currently enrolled in another clinical study or used any investigational drug or device within 28 days or 5*the half-life, whichever is longer preceding informed consent.
18. Known to be human immunodeficiency virus (HIV) positive at Screening.
19. Active viral hepatitis (B or C) as demonstrated by positive serology at Screening.
20. Has a current or prior diagnosis of narcolepsy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-08-12 (Actual)

PRIMARY OUTCOMES:
Ae: Cumulative Total (Unchanged) Amount of Lemborexant Excreted in Breast Milk Over the Entire Collection | 0-240 hours post-dose
Fraction (Percentage) of Dose Excreted in Breast Milk | 0-240 hours post-dose
  Fraction of dose excreted will be calculated as: Ae/Administered dose.
RID: Relative Infant Dose | 0-240 hours post-dose
  Relative infant dose is defined as the infant drug exposure via breast milk which is the body weight-adjusted percentage of maternal dose. Relative infant dose will be calculated by the formula: Daily infant dose milligram per kilogram (mg/kg)/maternal dose (mg/kg)*100, where estimated daily infant dose is as per the Food and Drug Administration (FDA) guidance (2019). Daily infant dose (mg/kg) = Ae/weight of infant.

SECONDARY OUTCOMES:
Number of Participants Reporting one or More Treatment-emergent Adverse Events (TEAEs) | Up to 215 days
Number of Participants Reporting one or More TEAEs Based on Severity | Up to 215 days
  All TEAEs will be graded on a 3-point scale (mild, moderate, and severe). The definitions are as follows: Mild (Discomfort noticed, but no disruption of normal daily activity); Moderate (Discomfort sufficient to reduce or affect normal daily activity); Severe (Incapacitating, with inability to work or to perform normal daily activity).
Number of Participants Reporting one or More TEAEs Based on Dose-relationship of Adverse Events (AEs) | Up to 215 days
Number of Participants With Clinically Significant Change in 12-lead Electrocardiogram (ECG) Findings | Up to 215 days
Number of Participants With Clinically Significant Change From Baseline in Vital Sign Values | Baseline up to 215 days
Number of Participants With Markedly Abnormal Change From Baseline in Laboratory Parameters | Baseline up to 215 days

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Phase 1 Clinic, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.

REFERENCES:
- [Derived] Rawal S, Brimhall D, Aluri J, Cheng JY, Hall N, Moline M. Lemborexant levels in breast milk after single doses in healthy, lactating women. Br J Clin Pharmacol. 2024 Jan;90(1):158-163. doi: 10.1111/bcp.15880. Epub 2023 Aug 23. PMID 37565541